CLINICAL TRIAL: NCT04275804
Title: Enhancement of Diabetic Foot Ulcer Healing Using Low-Magnitude High-Frequency Vibration Treatment - A Randomised Controlled Trial
Brief Title: Vibration Enhances Diabetic ULCER Healing
Acronym: VIBEDULCER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUHK
Record Dates: First submitted 2020-02-13; First posted 2020-02-19 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: Vibration; Whole Body Vibration; Low Magnitude High Frequency Vibration; Biophysical Intervention
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: conventional dressing (Active Comparator): Alternate day dressing in a designated clinic by a trained nurse specialized in wound care Dressing by a specialized wound-nurse is the current gold-stand of treatment for diabetic ulcers.
  Interventions: Other: Conventional Dressing
- Vibration group: conventional dressing and LMHFV (Experimental): Alternate day dressing in a designated clinic by a trained nurse specialized in wound care Alternate dat 20-week course of whole-body vibration therapy Alternate day 20min sessions on a self-designed vibration platform with low-magnitude high-frequency vibration (35Hz, 0.3g peak-to-peak displacement <0.1mm). Since the participants will return for dressing change on alternate days, the vibration group will also undergo the LMHFV on the same attendance.
  Interventions: Device: Low Magnitude High Frequence Vibration Platform

INTERVENTIONS:
Device: Low Magnitude High Frequence Vibration Platform — with low-magnitude high-frequency vibration (35Hz, 0.3g peak-to-peak displacement <0.1mm)
  Arms: Vibration group: conventional dressing and LMHFV
Other: Conventional Dressing — Alternate Day Dressing
  Arms: Control group: conventional dressing

SUMMARY:
Objectives:

Diabetes has a prevalence of 11.6% in China with diabetic foot ulcerations affecting over 30 million Chinese. 85% of these patients require amputation and 5-year mortality for diabetics is 70% when associated foot ulcers.

Clinical trials have shown that standing on whole-body vibration platforms, specifically low-magnitude high-frequency vibration (LMHFV); promotes angiogenesis, enhances muscle bulk and accelerates epithelization. Investigation on diabetic rats with foot wounds found accelerated wound healing, increased perfusion and upregulation of factors such as VEGF, PECAM-1 and PCNA.

Hypothesis:

The investigators postulate LMHFV will enhance diabetic foot ulcer healing.

Design and Subjects:

Prospective, single-centre, randomised control trial to treat 106 subjects with diabetic foot ulcers.

Interventions:

The intervention group will stand on LMHFV whole-body vibration platforms for 20min on alternate days for 20 weeks, together with conventional dressing by a trained wound-care nurse as in the control group.

Main Outcome Measures:

Ulcer size will be measured at multiple time points, the incidence of amputations/infections will be recorded, perfusion via ankle-brachial pressure index will be calculated and foot function via the foot and ankle outcome score will be analysed.

Data analysis:

Repeated measure of ANOVA to analyze time-point differences and student's t-test for same time-point comparison.

Expected Results:

This is the first clinical trial to investigate the effect of whole-body vibration on diabetic foot ulcers. It will show the investigators if the results from animal studies will translate into clinically significant results. If positive effects are established, whole-body vibration can be a valuable treatment regime to tackle diabetic foot ulcers.

DETAILED DESCRIPTION:
Plan of Investigation: (fig 04 in supplementary notes, CONSORT diagram)

Subjects:

Participants will be recruited from the patients in the Orthopaedic & Traumatology department at the Prince of Wales Hospital, the tertiary teaching hospital affiliated to CUHK.

Sample size: 106 subjects randomized 1:1 into the two treatment groups accounting for a dropout rate of 15%.

The sample size was calculated by using the primary endpoint of wound size in G*Power 3.1.9.4 (Germany). Using a 1:1 randomization ratio a type I error rate (a-level) of 0.05 and power of 0.95. Our vibration study of diabetic rat wounds showed an effect size d of 0.99. We estimate a tuned-down effect in human subjects, thus using an effect size of 0.7 we calculated that we should recruit 90 participants with 45 in each group. (22)

Methods:

Study Design:

Randomized Controlled Trial 1:1 randomization into control n=58 or intervention (Vibration) group n=58. Intervention

* Control group: conventional dressing
* Vibration group: conventional dressing + LMHFV

Data Analysis:

Randomisation performed using computer-generated randomization with a 1:1 allocation ratio using permuted block randomization to ensure similar numbers in the control and vibration group.

Compliance to intervention:

Conventional dressing: Each attendance to wound dressing will be recorded by the clinic nurse; those with <60% attendance to the wound clinic will be excluded.

LMHFV Vibration: each participant in the vibration intervention group will be assigned a personal 'smart card'. This smart card will record each utilization of the vibration platform to ensure compliance, those with <66% attendance will be excluded.

Repeated measures of ANOVA will be used to analyze the ulcer size groups and time points differences with be analyzed with post-hoc Bonferroni tests. Student's t-test for two independent samples will be used to compare groups of the same time point. Statistical analyses will be performed using IBM SPSS 25 (IBM, Armonk, NY, USA), and statistical significance was considered at p < 0.05.

ELIGIBILITY:
Inclusion criteria:

* >18 years old (legally able to self-sign consent)
* Able to stand independently
* Biochemically confirmed Diabetes with a fasting plasma glucose ≥ 7.0 mmol/L, or a random plasma glucose ≥ 11.1 mmol/L or hemoglobin A1c (HbA1c) level ≥ 6.5%
* Ulcers will be below the level of the malleoli, excluding those confined to the interdigital web space
* Cross-sectional area of the index ulcer should be 50- 1000 mm2
* Wagner stage 2-3
* Not active infection according to the Infectious Diseases Society of America guidelines

Exclusion criteria:

* Severe cognitive impairment or severe comorbidity, which may impair ability to adhere to intervention plan, e.g. severe dementia, poor cardiopulmonary reserve requiring home oxygen, daily hemodialysis etc.
* Evidence of active infection
* Recent revascularization procedure (<12 weeks)
* Recently received medication/intervention which might affect cell proliferation (eg chemotherapy, radiotherapy etc)
* Allergy to dressing, adhesives or antibiotics
* Incapable to understand the study protocol or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ulcer size | 0weeks, 2weeks, 8weeks, 14weeks, 20weeks, 56weeks
  • The baseline ulcer size will be measured at 0 weeks and a core interim measurement will be conducted at 20 weeks since 30% of ulcerations will heal at 20 weeks using conventional dressing. (13) A 1-year reassessment will help differentiate if the 20-week course of LMHFV therapy has created sustainable changes.

SECONDARY OUTCOMES:
Time (days) to healing | up to 56 weeks
  • The day of complete wound closure will be documented during their alternate day dressings in the designated clinic. The participant will still be reviewed at 20 weeks and 1 year for the primary outcome.
Incidence of amputation | up to 56 weeks
  • The reason and day of below knee/above knee amputation will be recorded. Details will be retrieved from the Clinical Management System, the centralized electronic healthcare system utilized by public hospitals in Hong Kong.
Incidence of secondary infection | up to 56 weeks
  • The number of hospitalized days and number of days of systemic antibiotic therapy will be documented. Details will be retrieved from the Clinical Management System, the centralized electronic healthcare system utilized by public hospitals in Hong Kong.
Perfusion | 0weeks, 20weeks
  • The measurement of the ABI will be standardized. (24) The subject will be at rest in supine position for 10mins, Doppler ultrasound to measure systolic blood pressure twice in the posterior tibial artery (If there is no obtainable signal in the posterior tibial artery, the dorsalis pedis will be used.), the average systolic blood pressure in the posterior tibial artery/dorsalis pedis divided by the higher of the SBP in the two arms will be used to calculate the ABI. (The higher SBP of the arm will be used in these calculations due to previous studies showing a strong association between peripheral arterial disease and subclavian stenosis)
Foot function | 0weeks, 20weeks
  • Foot function will be measured using the FAOS which is a variant of the KOOS specific for problems related to the foot and ankle region. The FAOS also has validated translations in English and Chinese; it is a questionnaire consisting of 5 Likert score subscales; Pain, Symptoms, ADL, Recreation and Foot related QOL. Answers are graded a score from 0-4 and a normalised score can be calculated for each subscale (100 is asymptomatic while 0 indicates extreme symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel KK Ling, MBChB, Principal Investigator — CUHK

IPD SHARING:
Plan to Share IPD: No